CLINICAL TRIAL: NCT05677854
Title: The Effect of Health Literacy Based Motivational Interviewing and Health Education on Nutrition and Physical Activity Behaviors of Adolescents
Brief Title: The Effect of Health Literacy Based Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşegül Akca (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Ayşegül Akca, Research Assistant, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022 - 042
Record Dates: First submitted 2022-12-29; First posted 2023-01-10 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-02

CONDITIONS: Health Literacy Level
Keywords: health literacy; motivational interview; health education; nutrition; physical activity; adolescent
MeSH Terms: conditions — Health Education; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational interview (Experimental): Motivational interviewing, consisting of 6 sessions with a one-week interval, was applied face to face to this intervention group. Each motivational interview lasted approximately 40 minutes.
  Interventions: Other: Health literacy based motivaonal interview
- Health education (Experimental): Health education consisting of 6 sessions, one week apart, was administered face to face to this intervention group. Each training session lasted approximately 40 minutes.
  Interventions: Other: Health literacy based health education
- Control (No Intervention): No intervention has been made.

INTERVENTIONS:
Other: Health literacy based motivaonal interview — Motivational interviewing technique was used based on health literacy.
  Arms: Motivational interview
Other: Health literacy based health education — Health education based on health literacy was used.
  Arms: Health education

SUMMARY:
It is important to adopt healthy lifestyle behaviors such as nutrition and physical activity in adolescence. Health literacy, which is the competence of adolescents to participate in their own health decisions and takes responsibility for health, needs to be developed. Developing healthy nutrition and physical activity behaviors with a focus on health literacy is important in terms of maintaining the desired behavior in adulthood. This study aims to examine the effects of health literacy-based motivational interviewing and health education on nutrition and exercise behaviors of adolescents. The research will be conducted with a single-blind randomized controlled experimental design. The population of the research consists of ninth-grade students. It is planned to include 72 people in the research sample according to the power analysis calculation. The research will be carried out with two intervention groups as motivational interview and health education and a control group.

ELIGIBILITY:
Inclusion Criteria:

* Continuing education in 9th grade
* Volunteering to participate in the research
* Permission by their families to participate in the research
* Being at a low or moderate level of health literacy according to the Health Literacy Scale for School-Age Children

Exclusion Criteria:

* Have a chronic illness
* Dieting within a program
* Doing regular physical activity
* Having a high level of health literacy according to the Health Literacy Scale for School-Age Children

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 63 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Health literacy level (Health Literacy Scale for School-Age Children) | before the implementation
  The level of health literacy was evaluated in three categories according to the score obtained: (10-25) points: low health literacy, (26-35) points: moderate health literacy and (36-40) points: high health literacy. By determining the health literacy level of the students, the intervention groups and the control group will be selected among the students with low and moderate health literacy levels.
Health literacy level (Health Literacy Scale for School-Age Children) | after the implementation
  The level of health literacy was evaluated in three categories according to the score obtained: (10-25) points: low health literacy, (26-35) points: moderate health literacy and (36-40) points: high health literacy. By determining the health literacy level of the students, the intervention groups and the control group will be selected among the students with low and moderate health literacy levels.
Health literacy level (Health Literacy Scale for School-Age Children) | three months after completion of the intervention
  The level of health literacy was evaluated in three categories according to the score obtained: (10-25) points: low health literacy, (26-35) points: moderate health literacy and (36-40) points: high health literacy.
Health literacy level (Health Literacy Scale for School-Age Children) | six months after completion of the intervention
  The level of health literacy was evaluated in three categories according to the score obtained: (10-25) points: low health literacy, (26-35) points: moderate health literacy and (36-40) points: high health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Çubuk/Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No